CLINICAL TRIAL: NCT00292760
Title: A Single-arm Phase II Study of Alemtuzumab in Combination With High-dose Methylprednisolone in CLL Patients With p53 Deletion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR2729; UKCLL 06 (CAM-PRED)
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Chronic Lymphocytic Leukaemia
MeSH Terms: conditions — Leukemia, B-Cell | interventions — Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab
Drug: Methyprednisolone

SUMMARY:
This is a phase II open label study for patients with p53-deleted CLL who require treatment. Both untreated and previously treated patients are eligible for study entry.

The trial consists of giving continuous alemtuzumab and cyclical high-dose methyl-prednisone.Alentuzumab is given intravenously during the first 4 weeks of treatment to ensure that adequate serum levels are achieved quickly. The drug will be administered daily during the first week, commencing at a dose of 3mg, and increasing to 10mg and then up to the target dose of 30mg as tolerated.Thereafter alemtuzumab will be given at a dose 30mg thrice weekly. From week 5, alemtuzumab will be given at the same dose but by the subcutaneous route of administration.

Methlyprednisolone will be given for 5 consecutive days at a daily dose of 1.0g/m2, starting on Day 1 and repeating the cycle every 28 days.

Treatment will be given for 16 weeks (i.e 4 cycles of methylprednisolone). Treatment will be discontinued if there is no response after 8 weeks, or if toxicity becomes unacceptable.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Written informed consent
* Confirmed diagnosis of CLL or SLL (small mature lymphocytes n blood, bone marrow or lymph nose expressing CD19, CD5, CD23, weakk CD79b, and weak clonally restricted immunoglobin light chain)
* p53 deletion by FISH in at least 20% of leukamia cells
* Treatment is indicated (Binet stage B or C, or stage A with a lyphocyte doubling time of less than 6 months, or disease-related symptoms or complications irrespective of clinical stage)
* WHO performance status 0, 1 or 2
* Both untreated and previously treated patients are eligible for study

Exclusion Criteria:

- Patients must have none of the following: Active infection Known HIV infection Past history of anaphylaxis following exposure to rat or mouse CDR-grafted humanised monoclonal antibodies Less than 3 weeks since prior chemotherapy Use of prior investigational agents within 6 weeks Pregnancy or lactation Uncontrolled diabetes mellitus Uncontrolled hypertension Active peptic ulcer disease Other severe concurrent diseases or mental disorders Serum urea or creatinine more than twice the upper limit of normal (unless due to uretic obstruction or renal infiltration by CLL/SLL) Serum bilirubin more than twice the upper limit of normal (unless due to haemlysis or liver infiltration with CLL/SLL) Persisting severe cytopenias due to previous therapy rather than disease (neutrophils <0.5 x 109/l or platelets <50 x 10/l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pettitt, Principal Investigator — Royal Liverpool University Hospital